CLINICAL TRIAL: NCT03965091
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Proof of Concept Study of the Efficacy and Safety of Fremanezumab for Treatment of Patients With Fibromyalgia
Brief Title: A Study to Test the Effectiveness and Safety of Fremanezumab on Participants With Fibromyalgia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Met pre-specified criteria for futility at interim analysis
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TV48125-PN-20028
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Results first posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — fremanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive placebo matching to fremanezumab SC on Days 1, 29, 57, and 85.
  Interventions: Drug: Placebo
- Fremanezumab Dose A (Experimental): Participants will receive fremanezumab SC on Days 1, 29, and 57 and placebo matched to fremanezumab SC on Day 85.
  Interventions: Drug: Fremanezumab
- Fremanezumab Dose B (Experimental): Participants will receive fremanezumab SC on Days 1, 29, and 57 and placebo matched to fremanezumab SC on Day 85.
  Interventions: Drug: Fremanezumab

INTERVENTIONS:
Drug: Fremanezumab — Fremanezumab will be administered per dose and schedule specified in the arm description.
  Arms: Fremanezumab Dose A; Fremanezumab Dose B
Drug: Placebo — Placebo matching to fremanezumab will be administered per schedule specified in the arm description.
  Arms: Placebo

SUMMARY:
The primary objective of the study is to estimate the treatment effect of fremanezumab administered subcutaneously (SC) in reducing pain in adult participants with fibromyalgia (FM). A secondary objective is to evaluate the effect of fremanezumab on other efficacy measures, including pain, quality of life, sleep, fatigue, improvement in health, physical functioning, and mood. Another secondary objective is to evaluate the safety and tolerability of fremanezumab administered SC in adult participants with FM.

The total duration of participant participation in the study is planned to be 21 weeks, consisting of a screening period of up to 5 weeks (ranging from 17 to 35 days), and a double-blind treatment period of 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* approved for study participation by the Fibromyalgia Eligibility Review Committee
* body mass index of 18.5 to 45 kilograms (kg)/square meter (m^2) and a body weight ≥45 kg
* agree to use only acetaminophen as rescue medication for FM-related pain (up to 1000 mg per dose and not to exceed 3000 mg/day for any indication throughout the study period)
* non-pharmacologic interventions (including normal daily exercise routines, chiropractic care, physical therapy, psychotherapy, and massage therapy) are unchanged for a minimum of 30 days prior to screening and will remain unchanged throughout the study
* agree to maintain a usual and unchanged physical exercise regimen
* must be of nonchildbearing potential or, defined as:

  * women surgically sterile by documented complete hysterectomy, bilateral oophorectomy, or
  * bitubal ligations or confirmed to be postmenopausal (at least 1 year since last menstrual period) and
  * menopausal women confirmed by a follicle-stimulating hormone >35 units (U)/liter (L)
  * men surgically sterile by documented vasectomy OR

If of childbearing potential, patients must meet any of the following criteria:

* must use highly effective contraception method with their partners during the entire study period and for 5 months after the last dose of the study drug.
* sexual abstinence is only considered a highly effective method if defined as refraining from heterosexual intercourse in the defined period.
* female participants of childbearing potential must have a negative serum beta-human chorionic gonadotropin (β-HCG) pregnancy test at screening (confirmed by urine dipstick β-HCG pregnancy test at baseline).

  * must agree not to participate in another interventional study from the screening period through the end of study (EOS) visit o Additional criteria apply, please contact the investigator for more information

Exclusion Criteria:

* unable or unwilling to discontinue/washout of prohibited medications
* ongoing pain that would confound or interfere with the assessment of the participant's FM pain or require excluded therapies during the participant's participation in this study.
* surgery planned during the study period
* receiving prophylactic treatment for migraine-related disorders, including topiramate, valproic acid, onabotulinumtoxinA, amitriptyline, and nortriptyline
* known history of clinically significant or unstable hematologic, cardiac, or thromboembolic events
* known history of suicide attempt, suicidal behavior, or suicidal ideation within the last 12 months
* lifetime history of any psychotic and/or bipolar disorder
* current, untreated, moderate or severe major depressive disorder and/or anxiety
* known history of hypersensitivity reactions to injected proteins, including monoclonal antibodies (mAbs) and animal venoms, or a history of Stevens-Johnson Syndrome/toxic epidermal necrolysis syndrome o Additional criteria apply, please contact the investigator for more information

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (49):
- United States (49):
  - Teva Investigational Site 14159, Birmingham, Alabama
  - Teva Investigational Site 14174, Huntsville, Alabama
  - Teva Investigational Site 14431, Mesa, Arizona
  - Teva Investigational Site 14166, Oceanside, California
  - Teva Investigational Site 14435, Panorama City, California
  - Teva Investigational Site 14168, Sacramento, California
  - Teva Investigational Site 14164, San Diego, California
  - Teva Investigational Site 14172, Torrance, California
  - Teva Investigational Site 14433, Stamford, Connecticut
  - Teva Investigational Site 14149, Ocala, Florida
  - Teva Investigational Site 14180, Oldsmar, Florida
  - Teva Investigational Site 14182, Plantation, Florida
  - Teva Investigational Site 14162, Tampa, Florida
  - Teva Investigational Site 14434, Marietta, Georgia
  - Teva Investigational Site 14148, Chicago, Illinois
  - Teva Investigational Site 14436, Flossmoor, Illinois
  - Teva Investigational Site 14155, Evansville, Indiana
  - Teva Investigational Site 14176, Overland Park, Kansas
  - Teva Investigational Site 14160, Wichita, Kansas
  - Teva Investigational Site 14429, Bowling Green, Kentucky
  - Teva Investigational Site 14147, North Dartmouth, Massachusetts
  - Teva Investigational Site 14157, Quincy, Massachusetts
  - Teva Investigational Site 14163, Ann Arbor, Michigan
  - Teva Investigational Site 14183, Hazelwood, Missouri
  - Teva Investigational Site 14170, O'Fallon, Missouri
  - Teva Investigational Site 14430, Springfield, Missouri
  - Teva Investigational Site 14165, Las Vegas, Nevada
  - Teva Investigational Site 14181, Albuquerque, New Mexico
  - Teva Investigational Site 14152, Raleigh, North Carolina
  - Teva Investigational Site 14185, Raleigh, North Carolina
  - Teva Investigational Site 14437, Salisbury, North Carolina
  - Teva Investigational Site 14167, Winston-Salem, North Carolina
  - Teva Investigational Site 14161, Fargo, North Dakota
  - Teva Investigational Site 14153, Cincinnati, Ohio
  - Teva Investigational Site 14432, Dayton, Ohio
  - Teva Investigational Site 14171, Portland, Oregon
  - Teva Investigational Site 14175, Salem, Oregon
  - Teva Investigational Site 14158, Allentown, Pennsylvania
  - Teva Investigational Site 14177, Duncansville, Pennsylvania
  - Teva Investigational Site 14156, Warwick, Rhode Island
  - Teva Investigational Site 14173, Knoxville, Tennessee
  - Teva Investigational Site 14150, Memphis, Tennessee
  - Teva Investigational Site 14151, Memphis, Tennessee
  - Teva Investigational Site 14178, Memphis, Tennessee
  - Teva Investigational Site 14184, Austin, Texas
  - Teva Investigational Site 14179, Dallas, Texas
  - Teva Investigational Site 14169, Salt Lake City, Utah
  - Teva Investigational Site 14146, Charlottesville, Virginia
  - Teva Investigational Site 14154, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo matched to fremanezumab subcutaneously (SC) on Days 1, 29, 57, and 85.
- Fremanezumab Dose A; Fremanezumab Dose B: Participants received fremanezumab SC on Days 1, 29, and 57 and placebo matched to fremanezumab SC on Day 85.
Period: Overall Study
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Started | 64 | 62 | 63
Received at Least 1 Dose of Study Drug | 64 | 62 | 63
Completed | 41 | 45 | 45
Not Completed | 23 | 17 | 18
Not completed — Adverse Event | 0 | 2 | 3
Not completed — Withdrawal by Subject | 11 | 3 | 5
Not completed — Non-compliance with study drug | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Other than specified | 9 | 11 | 8

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set included all randomized participants.
Groups:
- Placebo: Participants received placebo matched to fremanezumab SC on Days 1, 29, 57, and 85.
- Total: Total of all reporting groups
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B | Total
Number analyzed (Participants) | 64 | 62 | 63 | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (11.54) | 52.3 (11.75) | 52.2 (12.59) | 51.9 (11.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 59 | 59 | 178
  Male | 4 | 3 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 9 | 7 | 22
  Not Hispanic or Latino | 58 | 53 | 55 | 166
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 58 | 50 | 54 | 162
  Race: Black or African American | 5 | 9 | 5 | 19
  Race: Asian | 0 | 0 | 2 | 2
  Race: American Indian or Alaska Native | 0 | 1 | 1 | 2
  Race: Other | 1 | 2 | 1 | 4
Weekly Average of the Daily Average Pain Intensity-Numerical Rating Scale (PI-NRS) Score [Mean (Standard Deviation); unit: units on a scale] — The PI-NRS is an 11-point pain intensity numerical rating scale where 0=no pain and 10=worst possible pain; higher scores indicating more pain. Weekly average of the daily average PI-NRS pain score over the past 24 hours was derived using formula: Summation of non-missing efficacy variable in an analysis week divided by the number of days with non-missing efficacy variable in the analysis week.
  units on a scale | 5.6 (1.05) | 5.8 (1.03) | 6.0 (1.11) | 5.8 (1.07)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Weekly Average of the Daily Average Pain Intensity-Numerical Rating Scale (PI-NRS) Score Over the Past 24 Hours at Week 12
Description: The PI-NRS is an 11-point pain intensity numerical rating scale where 0=no pain and 10=worst possible pain; higher scores indicating more pain. Weekly average of the daily average PI-NRS pain score over the past 24 hours was derived using formula: Summation of non-missing efficacy variable in an analysis week divided by the number of days with non-missing efficacy variable in the analysis week. Baseline was defined as the last 14 days before the first dose of study drug.
Time Frame: Baseline, Week 12
Population: Modified intent-to-treat (mITT) analysis set included all randomized participants who received at least 1 dose of study drug and at least 1 postbaseline entry of daily average pain intensity using the PI-NRS. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 46 | 52 | 50
units on a scale | -1.5 (1.79) | -1.2 (1.58) | -1.3 (1.61)
Statistical Analysis 1: Comparison: Placebo vs Fremanezumab Dose A; Analysis was performed using a Mixed Model Repeated Measures (MMRM) model with change from baseline in the weekly average of the daily average PI-NRS score over the past 24 hours at weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 as the dependent variable, sex, age group at FM onset, week, treatment, and treatment-by-week interaction as fixed factors, and baseline average of the daily average PI-NRS score as a covariate; Test type: Other; p = 0.7963, Mixed Models Analysis; Least square (LS) mean difference = 0.1, 95% CI 2-sided [-0.46 to 0.60], Standard Error of Mean 0.27
Statistical Analysis 2: Comparison: Placebo vs Fremanezumab Dose B; Analysis was performed using an MMRM model with change from baseline in the weekly average of the daily average PI-NRS score over the past 24 hours at weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 as the dependent variable, sex, age group at FM onset, week, treatment, and treatment-by-week interaction as fixed factors, and baseline average of the daily average PI-NRS score as a covariate; Test type: Other; p = 0.8629, Mixed Models Analysis; LS mean difference = 0.0, 95% CI 2-sided [-0.48 to 0.58], Standard Error of Mean 0.27

2. Secondary Outcome: Change From Baseline in the Individual Components of the Fibromyalgia Impact Questionnaire Revised (FIQR) Score: Symptom Subscore, Impact Subscore, and Functional Subscore at Week 12
Description: The FIQR is a commonly used instrument in the evaluation of fibromyalgia participants. It contains 21 questions in 3 domains: function (9 questions), overall impact (2 questions), and symptoms (10 questions). Questions are graded on a 0 to 10 numeric scale with 10 being the worst. All questions are framed in the context of the last 7 days. The sub-total score for each domain is the summation of scores in the domain. The function sub-total score ranges from 0 (better) to 90 (worst), with a lower score indicating better (higher) function; overall impact sub-total score ranges from 0 to 20, with a lower score indicating better (lower) impact; the symptoms sub-total score ranges from 0 to 100, with a lower score indicating a better (lower) level of symptoms. Baseline was defined as the last 14 days before the first dose of study drug.
Time Frame: Baseline, Week 12
Population: mITT analysis set included all randomized participants who received at least 1 dose of study drug and at least 1 postbaseline entry of daily average pain intensity using the PI-NRS. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 43 | 45 | 46
units on a scale
  Change at Week 12 in Symptoms Subscore | -9.1 (13.99) | -4.0 (13.76) | -8.1 (15.19)
  Change at Week 12 in Impact Subscore | -2.0 (4.60) | -1.6 (5.00) | -2.2 (4.27)
  Change at Week 12 in Functional Subscore | -9.5 (16.26) | -4.7 (18.54) | -6.7 (13.35)

3. Secondary Outcome: Responder Rate of the Patient Global Impression of Change (PGIC) Rating: Number of Participants Who Were Much Improved or Very Much Improved at Week 12
Description: The PGIC scale evaluates all aspects of participants' health and assesses if there has been an improvement or decline in clinical status since the start of the study. Participants recorded responses to the PGIC scale at Week 12. Improvement was recorded on a 7-point scale, with 1 = very much improved, 2 = Much Improved, 3 = Minimally Improved, 4 = No Change, 5 = Minimally Worse, 6 = Much Worse, and 7 = Very Much Worse. Scale "much improved" or "very much improved" were considered improved.
Time Frame: Week 12
Population: mITT analysis set included all randomized participants who received at least 1 dose of study drug and at least 1 postbaseline entry of daily average pain intensity using the PI-NRS.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 64 | 62 | 63
Participants | 14 | 12 | 11

4. Secondary Outcome: Number of Participants Who Experienced ≥30% Reduction From Baseline in Weekly Average of Daily Average PI-NRS Score at Week 12
Description: The PI-NRS is an 11-point pain intensity numerical rating scale where 0=no pain and 10=worst possible pain; higher scores indication more pain. Weekly average of the daily average PI-NRS pain score over the past 24 hours was derived using formula: Summation of non-missing efficacy variable in an analysis week divided by the number of days with non-missing efficacy variable in the analysis week.
Time Frame: Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 46 | 52 | 50
Participants | 19 | 18 | 18

5. Secondary Outcome: Number of Participants Who Experienced ≥50% Reduction From Baseline in Weekly Average of Daily Average PI-NRS Score at Week 12
Description: as for outcome 4
Time Frame: Week 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 46 | 52 | 50
Participants | 11 | 6 | 8

6. Secondary Outcome: Change From Baseline in the Weekly Average of Daily Worst PI-NRS Score Over Past 24 Hours at Week 12
Description: The PI-NRS is an 11-point pain intensity numerical rating scale where 0=no pain and 10=worst possible pain; higher scores indication more pain. Weekly average of the daily worst PI-NRS pain score over the past 24 hours was derived using formula: Summation of non-missing efficacy variable in an analysis week divided by the number of days with non-missing efficacy variable in the analysis week. Baseline was defined as the last 14 days before the first dose of study drug.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 46 | 52 | 50
units on a scale | -1.6 (2.00) | -1.4 (1.54) | -1.3 (1.80)

7. Secondary Outcome: Change From Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short Form (SF) 8a T-score at Week 12
Description: The PROMIS SF8a scale contains 8 items and assesses sleep disturbance over the past 7 days. One item assessing overall sleep quality use a scale of very poor, poor, fair, good, or very good. Other 7 items use a scale of not at all, a little bit, somewhat, quite a bit, or very much. Each item of the PROMIS sleep disturbance SF8a is on 5-point scales (1 to 5), with 1 for the lowest sleep disturbance and 5 for the highest sleep disturbance. The total score ranging from 8 (lowest sleep disturbance) to 40 (highest sleep disturbance) was calculated as the summation of 8 non-missing scores. T-score was calculated from the total raw score using the scoring table (PROMIS-Sleep Disturbance Scoring Manual) with a mean of 50 and a standard deviation of 10. Possible range for T-score is 30 to 80, with higher scores indicating greater severity of sleep impairment.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 43 | 46 | 42
T-score | -4.7 (8.39) | -2.6 (8.31) | -3.1 (6.86)

8. Secondary Outcome: Change From Baseline in the PROMIS Physical Function SF 12a Scale Score at Week 12
Description: The PROMIS physical function scale measures self-reported capability. This includes the functioning of one's upper extremities (dexterity), lower extremities (walking or mobility), and central regions (neck, back), as well as instrumental activities of daily living, such as running errands over the past 7 days. A single physical function capability score is obtained from a SF. The PROMIS physical function SF12a scale contains 12 items with 5-point scales (1 [not at all] to 5 [very much]) for each item with a total score ranging from 12 (poor physical function) to 60 (better physical function). A higher score indicates greater level of physical capability. Total raw score was calculated as the summation of 12 non-missing scores for participants who can walk 25 feet or summation of 6 non-missing scores for participants who cannot walk for 25 feet. The calculated total raw score was converted into scale score using the scoring tables (PROMIS-Physical Function Scoring Manual).
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 43 | 45 | 46
units on a scale | 1.8 (3.67) | 0.7 (4.28) | 1.0 (3.59)

9. Secondary Outcome: Change From Baseline in the PROMIS Fatigue SF 8a T-Score at Week 12
Description: The PROMIS Fatigue SF8a contains 8 items with 5-point scales (1 [never] to 5 [always]) for each item over the past 7 days. The total raw score ranges from 8 (lowest level of fatigue) to 40 (highest level of fatigue) was calculated as the summation of 8 non-missing scores. T-score was calculated from the total raw score using the scoring table (PROMIS-Fatigue Scoring Manual) with a mean of 50 and a standard deviation of 10; scores higher than 50 indicate greater fatigue compared to the reference population.
Time Frame: Baseline, Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 43 | 45 | 45
T-score | -3.9 (8.61) | -3.3 (6.92) | -3.3 (7.97)

10. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse events (SAEs) were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. Any AE occurring on or after the first dose of study drug is considered a treatment-emergent AE (TEAE). A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Baseline up to Week 16
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 64 | 62 | 63
Participants | 34 | 30 | 29

11. Secondary Outcome: Number of Participants With at Least 1 Potentially Clinically Significant Abnormal Serum Chemistry Value
Description: Potentially clinically significant serum chemistry abnormalities included: Blood urea nitrogen ≥10.71 millimoles (mmol)/liter (L) and Gamma-glutamyl transpeptidase (GGT) ≥3 * upper limit of normal (ULN).
Time Frame: Baseline up to Week 16
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 61 | 60 | 62
Participants | 2 | 2 | 1

12. Secondary Outcome: Number of Participants With at Least 1 Potentially Clinically Significant Abnormal Hematology Value
Description: Potentially clinically significant hematological abnormalities included: White blood cells (WBCs) count ≤3.0 * 10^9/L; Hemoglobin ≤95 grams (g)/L in females; Hematocrit <0.32 L/L in females; Platelets ≥700 * 10^9/L; and Eosinophils/Leukocytes ≥10%.
Time Frame: Baseline up to Week 16
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 61 | 60 | 62
Participants | 4 | 3 | 7

13. Secondary Outcome: Number of Participants With at Least 1 Potentially Clinically Significant Urinalysis Abnormalities
Time Frame: Baseline up to Week 16
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 64 | 62 | 63
Participants | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With at Least 1 Clinically Significant Abnormal Vital Signs Value
Description: Clinically significant vital signs abnormalities included: Systolic blood pressure (BP): ≤90 millimeters of mercury (mmHg) and decrease from baseline of 20 mm Hg; Diastolic BP: ≥105 mmHg and increase from baseline of ≥15 mmHg or ≤50 mmHg and decrease from baseline of ≥15 mmHg.
Time Frame: Baseline up to Week 16
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 62 | 60 | 62
Participants | 1 | 2 | 0

15. Secondary Outcome: Number of Participants With at Least 1 Physical Examination Abnormal Finding
Description: Physical examination included: General appearance, HEENT (head, ears, eyes, nose, and throat examination), chest and lungs, heart, cardiovascular, abdomen, musculoskeletal, skin, lymph nodes, neurological, and extremities/back.
Time Frame: Baseline up to Week 16
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 64 | 62 | 63
Participants | 24 | 25 | 28

16. Secondary Outcome: Number of Participants With Shift From Baseline to Endpoint in Electrocardiogram (ECG) Parameters
Description: The number of participants with a difference (shift) from baseline in any of the following ECG parameters is reported by group: heart rate, PR interval, QRS interval, RR interval, QT interval corrected usingthe Fridericia formula (QTcF) and QT interval corrected using the Bazett's formula (QTcB). Shifts represented as Baseline - endpoint value (last observed post-baseline value).
Time Frame: Baseline to Week 16
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug. Here, 'Overall number of participants analyzed' = participants with both baseline and postbaseline ECG value.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 58 | 55 | 59
Participants
  Normal - Normal | 39 | 36 | 34
  Normal - Abnormal, not clinically significant | 9 | 11 | 6
  Normal - Abnormal, clinically significant | 0 | 0 | 1
  Abnormal - Normal | 4 | 2 | 5
  Abnormal - Abnormal, not clinically significant | 6 | 6 | 12
  Abnormal - Abnormal, clinically significant | 0 | 0 | 1

17. Secondary Outcome: Number of Participants With at Least 1 Injection Site AE
Description: Injection site AEs included injection site pain, injection site erythema, injection site induration, injection site pruritus, injection site bruising, injection site nodule, injection site swelling, and injection site warmth.
Time Frame: Baseline up to Week 16
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 64 | 62 | 63
Participants | 5 | 8 | 7

18. Secondary Outcome: Number of Participants With Hypersensitivity/Anaphylaxis Reactions
Time Frame: Baseline up to Week 16
Population: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 64 | 62 | 63
Participants | 0 | 1 | 0

19. Secondary Outcome: Time to Withdrawal of Treatment Due to Lack of Efficacy
Time Frame: Baseline up to Week 16
Population: mITT analysis set included all randomized participants who received at least 1 dose of study drug and at least 1 postbaseline entry of daily average pain intensity using the PI-NRS. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. There were no participants with evaluable data in the Fremanezumab Dose B arm.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 2 | 1 | 0
weeks | NA [NA to NA] — Due to small number of participants who withdrew treatment due to lack of efficacy, median and 95% confidence interval (CI) could not be calculated. | NA [NA to NA] — Due to small number of participants who withdrew treatment due to lack of efficacy, median and 95% CI could not be calculated. |

20. Secondary Outcome: Time to Withdrawal of Treatment Due to AEs
Time Frame: Baseline up to Week 16
Population: mITT analysis set included all randomized participants who received at least 1 dose of study drug and at least 1 postbaseline entry of daily average pain intensity using the PI-NRS. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure. There were no participants with evaluable data in the Placebo arm.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
Number analyzed (Participants) | 0 | 2 | 3
weeks |  | NA [NA to NA] — Due to small number of participants who withdrew treatment due to AEs, median and 95% CI could not be calculated. | NA [NA to NA] — Due to small number of participants who withdrew treatment due to AEs, median and 95% CI could not be calculated.

ADVERSE EVENTS:
Time Frame: Baseline up to Week 16
Description: Safety analysis set included all randomized participants who received at least 1 dose of study drug.
Arm/Group | Placebo | Fremanezumab Dose A | Fremanezumab Dose B
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/62 | 0/63
Serious Adverse Events (participants affected / at risk) | 1/64 | 1/62 | 1/63
Other Adverse Events (participants affected / at risk) | 8/64 | 14/62 | 10/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=64) | Fremanezumab Dose A (N=62) | Fremanezumab Dose B (N=63)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=64) | Fremanezumab Dose A (N=62) | Fremanezumab Dose B (N=63)
Nausea (Gastrointestinal disorders) | 1 (2) | 4 (4) | 1 (1)
Injection site erythema (General disorders) | 3 (7) | 6 (14) | 3 (7)
Injection site induration (General disorders) | 1 (2) | 1 (3) | 5 (23)
Injection site pain (General disorders) | 4 (10) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (4) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2021-08-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT03965091/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT03965091/SAP_001.pdf